CLINICAL TRIAL: NCT05156125
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Clinical Efficacy and Safety of VTX002 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: VTX002 Versus Placebo for the Treatment of Moderately to Severely Active Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oppilan Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX002-201
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Colitis, Ulcerative
Keywords: S1P; sphingosine 1 phosphate receptor;; Ventyx; Oppilan;; moderate or severe ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will employ a double-blind design. Subjects, Investigators, study center staff, persons performing the assessments, central endoscopy readers and the Sponsor are to remain blinded to the identity of the Induction Period treatment from the time of randomization until the interim database lock for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VTX002 Dose A (Experimental): VTX002 Dose A tablet administered orally once daily
  Interventions: Drug: VTX002
- VTX002 Dose B (Experimental): VTX002 Dose B tablet administered orally once daily
  Interventions: Drug: VTX002
- Placebo (Placebo Comparator): Placebo tablet administered orally once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VTX002 — Dose A tablet administered orally once daily
  Other Names: OPL-002
  Arms: VTX002 Dose A
Drug: VTX002 — Dose B Tablet administered orally once daily
  Other Names: OPL-002
  Arms: VTX002 Dose B
Drug: Placebo — Placebo Tablet for VTX002 administered orally once daily
  Arms: Placebo

SUMMARY:
This is a study to understand if taking VTX002 daily as a tablet orally is safe and effective in participants diagnosed with moderate to severe ulcerative colitis (UC). Approximately 189 participants will take VTX002 Dose A, VTX002 Dose B, or matching placebo, once daily.

The study consists of a 28-day Screening Period (to see if a participant qualifies for the study), a 13-week double-blind period (a participant receives either active Dose A, Dose B or Placebo), a Long-Term Extension (LTE) Treatment Period of up to 39 weeks, an Open-Label Extension (OLE) Treatment Period of up to 143 weeks, and a 2-week Follow-Up Period. The maximal duration of treatment including the Induction Period, LTE and OLE will be 36 months.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of VTX002 in subjects with moderately to severely active UC following daily oral administration of VTX002 as a tablet. Approximately 189 eligible subjects will be randomized in a 1:1:1 ratio to receive VTX002 Dose A, VTX002 Dose B, or matching placebo, once daily (approximately 63 subjects per treatment group).

The study consists of a 28-day Screening Period, a 13-week double-blind Induction Treatment Period (including 7 days of titration followed by 12 weeks of treatment at the assigned dose), a Long-Term Extension (LTE) Treatment Period of up to 39 weeks, an Open-Label Extension (OLE) Treatment Period of up to 143 weeks, and a 2-week Follow-Up Period. The maximal duration of treatment including the Induction Period, LTE and OLE will be 36 months.

Objectives Primary Objective

• Assess the efficacy of VTX002 when administered for 13 weeks on clinical remission

Secondary Objectives

* Assess the efficacy of VTX002 when administered for 13 weeks on endoscopic changes, symptomatic response and remission, histology, and mucosal healing
* Assess the safety and tolerability of VTX002
* Assess the pharmacokinetics (PK) of VTX002

Long-Term and Open-Label Extension Objectives

* Assess the efficacy of VTX002 through the LTE and OLE Treatment Periods on endoscopic changes, symptomatic response and remission, histology, and mucosal healing
* Assess the safety of VTX002 through the LTE and OLE Treatment Periods

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with UC ≥ 3 months prior to Screening.
* Active UC confirmed by endoscopy

Exclusion Criteria:

* Severe extensive colitis
* Diagnosis of Crohn's disease (CD) or indeterminate colitis or the presence or history of a fistula consistent with CD
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2026-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Naik, PhD, Study Director — Ventyx Biosciences, Inc
Locations (77):
- United States (19):
  - Local Site # 840030, Garden Grove, California
  - Local Site # 840026, Lancaster, California
  - Local Site # 840040, San Diego, California
  - Local Site # 840001, Ventura, California
  - Local Site # 840049, Kissimmee, Florida
  - Local Site # 840006, Miami, Florida
  - Local Site # 840018, Atlanta, Georgia
  - Local Site # 840046, New Albany, Indiana
  - Local Site # 840042, Shreveport, Louisiana
  - Local Site # 840044, Ypsilanti, Michigan
  - Local Site # 840043, Dayton, Ohio
  - Local Site # 840010, Oklahoma City, Oklahoma
  - Local Site # 840045, Myrtle Beach, South Carolina
  - Local Site # 840013, Garland, Texas
  - Local Site # 8400039, Lubbock, Texas
  - Local Site # 840033, McAllen, Texas
  - Local Site # 840007, San Marcos, Texas
  - Local Site # 840016, Southlake, Texas
  - Local Site # 840028, Tyler, Texas
- Bulgaria (2):
  - Local Site # 100002, Rousse
  - Local Site # 100005, Rousse
- Czechia (3):
  - Local Site # 203002, Hradec Králové
  - Local Site # 203001, Slaný
  - Local Site # 203004, Ústí nad Labem
- France (3):
  - Local Site # 250004, Caen
  - Local Site # 250001, Nantes
  - Local Site # 250003, Vandœuvre-lès-Nancy
- Georgia (6):
  - Local Site # 268001, Tbilisi
  - Local Site # 268002, Tbilisi
  - Local Site # 268003, Tbilisi
  - Local Site # 268004, Tbilisi
  - Local Site # 268005, Tbilisi
  - Local Site # 268006, Tbilisi
- Germany (5):
  - Local Site # 276005, Berlin
  - Local Site # 276008, Brandenburg
  - Local Site # 276007, Duisburg
  - Local Site # 276009, Halle
  - Local Site # 276003, Nordhausen
- Hungary (4):
  - Local Site # 348004, Békéscsaba
  - Local Site # 348001, Budapest
  - Local Site # 348003, Budapest
  - Local Site # 348002, Székesfehérvár
- India (3):
  - Local Site # 356001, Ahmedabad
  - Local Site # 356003, Jaipur
  - Local Site # 356005, Sūrat
- Italy (5):
  - Local Site # 380009, Milan
  - Local Site # 380001, Negrar
  - Local Site # 380004, Pavia
  - Local Site # 380008, Rome
  - Local Site # 380002, San Giovanni Rotondo
- Lithuania (2):
  - Local Site # 440002, Panevezys
  - Local Site # 440001, Vilnius
- Poland (15):
  - Local Site # 616010, Bydgoszcz
  - Local Site # 616012, Jelenia Góra
  - Local Site # 616001, Lodz
  - Local Site # 616017, Lodz
  - Local Site # 616015, Lublin
  - Local Site # 616004, Oświęcim
  - Local Site # 616011, Piotrkow Trybunalski
  - Local Site # 616008, Poznan
  - Local Site # 616014, Rzeszów
  - Local Site # 616007, Sosnowiec
  - Local Site # 616003, Warsaw
  - Local Site # 616006, Warsaw
  - Local Site # 616002, Wroclaw
  - Local Site # 616009, Wroclaw
  - Local Site # 616013, Wroclaw
- Serbia (4):
  - Local Site # 688002, Belgrade
  - Local Site # 688003, Belgrade
  - Local Site # 688004, Belgrade
  - Local Site # 688001, Zrenjanin
- Slovakia (3):
  - Local Site # 703001, Košice
  - Local Site # 703003, Prešov
  - Local Site # 703002, Šahy
- South Korea (3):
  - Local Site # 410003, Daegu
  - Local Site # 410002, Seoul
  - Local Site # 410004, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sands BE, Panaccione R, D'Haens G, Schreiber S, Jairath V, DuVall A, Kierkus J, Walczak M, Naik S, Gilder K, Lindstrom B, Ogilvie K, Sandborn WJ, Vermeire S, Rubin DT, Peyrin-Biroulet L, Danese S. Tamuzimod in patients with moderately-to-severely active ulcerative colitis: a multicentre, double-blind, randomised, placebo-controlled, phase 2 induction trial. Lancet Gastroenterol Hepatol. 2025 Mar;10(3):210-221. doi: 10.1016/S2468-1253(24)00386-8. Epub 2025 Jan 7. PMID 39793589

RESULTS

PARTICIPANT FLOW:
Groups:
- VTX002 60 mg Once Daily: VTX002 60 mg tablet administered orally once daily
- VTX002 30 mg Once Daily: VTX002 30 mg tablet administered orally once daily
- Placebo Once Daily: Placebo tablet administered orally once daily
Period: Overall Study
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Started | 70 | 73 | 70
Entered Long-Term Extension Following Induction | 29 | 34 | 22
Entered Open-Label Extension Following Induction | 37 | 36 | 42
Did Not Enter Long-Term or Open-Label Extension Following Induction | 1 | 0 | 2
Completed (Completed Induction Treatment Period; participants who completed this study period could have entered the Long-Term Extension or Open-Label Extension Periods) | 67 | 70 | 66
Not Completed | 3 | 3 | 4
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Non-compliance | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Consists of all randomized participants receiving at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily | Total
Number analyzed (Participants) | 70 | 73 | 70 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (13.81) | 42.3 (15.01) | 40.1 (13.78) | 40.6 (14.21)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 | 49 | 41 | 46 | 136
  45 to 65 | 18 | 27 | 21 | 66
  >65 | 3 | 5 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 26 | 32 | 97
  Male | 31 | 47 | 38 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 3 | 13
  Not Hispanic or Latino | 67 | 66 | 66 | 199
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 4 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 60 | 67 | 63 | 190
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission at 13 Weeks
Description: The percentage of participants with clinical remission at Week 13. Clinical remission was based on the modified Mayo score (MMS), which is a composite score of participant-reported symptoms and endoscopies which were assessed by a central reader. Clinical remission was defined as stool frequency (SF) subscore = 0 or 1, rectal bleeding (RB) subscore = 0, and endoscopic subscore (ES) ≤ 1 (excluding friability). Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Day 1 of Induction treatment period to Week 13
Population: Full Analysis Set - Baseline Modified Mayo Score 5-9
Measure: Count of Participants; unit: Participants
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 68 | 71 | 70
Participants | 19 | 17 | 8
Statistical Analysis 1: Comparison: VTX002 60 mg Once Daily vs Placebo Once Daily; At 13 weeks; Test type: Superiority; p = 0.0184, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.1, 95% CI 2-sided [2.58 to 29.05]
Statistical Analysis 2: Comparison: VTX002 30 mg Once Daily vs Placebo Once Daily; At 13 weeks; Test type: Superiority; p = 0.0410, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.1, 95% CI 2-sided [-0.03 to 25.58]

2. Secondary Outcome: Endoscopic Improvement at Week 13
Description: The percentage of participants with endoscopic improvement at Week 13. Endoscopic improvement was assessed from endoscopies assessed by a central reader. Endoscopic improvement was defined as ES ≤ 1 (excluding friability). The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease).
Time Frame: Day 1 of Induction Treatment Period to Week 13
Population: Full Analysis Set - Baseline MMS 5 to 9
Measure: Count of Participants; unit: Participants
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 68 | 71 | 70
Participants | 25 | 23 | 11
Statistical Analysis 1: Comparison: VTX002 60 mg Once Daily vs Placebo Once Daily; At 13 weeks; Test type: Superiority; p = 0.0070, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.6, 95% CI 2-sided [5.73 to 34.42]
Statistical Analysis 2: Comparison: VTX002 30 mg Once Daily vs Placebo Once Daily; At Week 13; Test type: Superiority; p = 0.0162, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.3, 95% CI 2-sided [2.75 to 30.67]

3. Secondary Outcome: Symptomatic Remission at Week 13
Description: The percentage of participants with symptomatic remission at Week 13. Symptomatic remission was measured using participant-reported symptoms and was defined as SF subscore = 0 or 1 and RB subscore = 0. The SF subscore ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB subscore ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicate more severe disease.
Time Frame: Day 1 of Induction Treatment Period to Week 13
Population: Full analysis set - Baseline MMS 5 to 9
Measure: Count of Participants; unit: Participants
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 68 | 71 | 70
Participants | 29 | 29 | 18
Statistical Analysis 1: Comparison: VTX002 60 mg Once Daily vs Placebo Once Daily; Test type: Superiority; p = 0.0448, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.5, 95% CI 2-sided [0.65 to 31.37]
Statistical Analysis 2: Comparison: VTX002 30 mg Once Daily vs Placebo Once Daily; At Week 13; Test type: Superiority; p = 0.0417, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.0, 95% CI 2-sided [0.23 to 30.58]

4. Secondary Outcome: Histologic Remission at Week 13
Description: The percentage of participants with histologic remission at Week 13. Histologic remission was assessed using the Geboes Index score and defined for this outcome measure as a Geboes score < 2.0. The Geboes score grading system is a validated score for evaluating histologic disease activity in ulcerative colitis and is graded on a scale of 0 to 5. A higher Geboes score indicates more severe disease.
Time Frame: Day 1 of Induction Treatment Period to Week 13
Population: Full analysis set - Baseline MMS 5 to 9
Measure: Count of Participants; unit: Participants
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 68 | 71 | 70
Participants | 13 | 20 | 5
Statistical Analysis 1: Comparison: VTX002 60 mg Once Daily vs Placebo Once Daily; Test type: Superiority; p = 0.0499, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.5, 95% CI 2-sided [-0.99 to 23.38]
Statistical Analysis 2: Comparison: VTX002 30 mg Once Daily vs Placebo Once Daily; At Week 13; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.4, 95% CI 2-sided [7.94 to 33.53]

5. Secondary Outcome: Endoscopic Improvement-Histologic Remission at Week 13
Description: The percentage of participants with endoscopic improvement-histologic remission at Week 13. This outcome measure was assessed by endoscopic histologic scores and defined as ES ≤ 1 (excluding friability) and a Geboes Index score < 2.0. The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease). The Geboes score grading system is a validated score for evaluating histologic disease activity in ulcerative colitis and is graded on a scale of 0 to 5. A higher Geboes score indicates more severe disease.
Time Frame: Day 1 of Induction Treatment Period to Week 13
Population: Full Analysis Set - Baseline MMS 5 to 9
Measure: Count of Participants; unit: Participants
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
Number analyzed (Participants) | 68 | 71 | 70
Participants | 7 | 14 | 0
Statistical Analysis 1: Comparison: VTX002 60 mg Once Daily vs Placebo Once Daily; At Week 13; Test type: Superiority; p = 0.0072, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: VTX002 30 mg Once Daily vs Placebo Once Daily; At Week 13; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: PK of VTX002
Description: Plasma concentrations of VTX002 in samples obtained predose at Weeks 1, 4, 8, and 13 in the Induction Treatment Period
Time Frame: Weeks 1, 4, 8, and 13 of the Induction Treatment Period
Population: The Pharmacokinetics Set consisted of all participants who received VTX002 and had at least 1 measured concentration at a scheduled PK timepoint after start of dosing for VTX002.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily
Number analyzed (Participants) | 70 | 73
ng/mL
  Week 1 | 640.8 (378.77) | 363.2 (237.79)
  Week 4 | 911.5 (777.40) | 374.7 (242.93)
  Week 8 | 935.1 (718.16) | 393.2 (251.98)
  Week 13 | 1050 (930.15) | 444.2 (341.13)

ADVERSE EVENTS:
Time Frame: From the signing of the Informed Consent Form through 30 days after the last study treatment, up to 13 weeks in the Induction Treatment Period.
Groups:
- Placebo Once Daily: Placebo tablet for VTX002 administered orally once daily
Arm/Group | VTX002 60 mg Once Daily | VTX002 30 mg Once Daily | Placebo Once Daily
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/73 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/70 | 2/73 | 0/70
Other Adverse Events (participants affected / at risk) | 10/70 | 10/73 | 9/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VTX002 60 mg Once Daily (N=70) | VTX002 30 mg Once Daily (N=73) | Placebo Once Daily (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VTX002 60 mg Once Daily (N=70) | VTX002 30 mg Once Daily (N=73) | Placebo Once Daily (N=70)
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 1
Headache (Nervous system disorders) | 4 | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT05156125/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT05156125/SAP_001.pdf